CLINICAL TRIAL: NCT06966947
Title: The Positive Impact of Risk Early Warning Management on Postoperative Rehabilitation Quality and Incidence of Delirium in Patients With Hip Fractures
Brief Title: Risk Early Warning Management for Postoperative Hip Fracture Rehabilitation and Delirium Prevention in Elderly Patients
Status: Completed | Type: Observational
Sponsor: People's Hospital Affiliated to Hubei University of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PeoplesHospitalHubei
Record Dates: First submitted 2025-04-09; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hip Fractures (ICD-10 72.01-72.2)
Keywords: Risk early warning management; Hip fracture rehabilitation; Postoperative delirium prevention; Proximal femoral nail (PFN) surgery; Elderly orthopedic patients; Blood coagulation function; Self-care ability; Retrospective cohort study
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Risk Early Warning Perioperative Management: Participants in this arm received a structured risk early warning management intervention during the perioperative period. The intervention included the establishment of a dedicated nursing team, systematic evaluation of vital signs (heart rate, respiratory rate, blood pressure, temperature, and consciousness), and scoring of patient condition based on a predefined risk assessment table.
  Based on the risk score, patients received tiered monitoring and intervention:
  Score 0-4: Routine care and monitoring
  Score 5-7 or single item score = 3: Intensive monitoring every 4 hours and physician notification
  Score ≥7: Continuous monitoring, immediate physician arrival, and bedside emergency preparedness This strategy aimed to detect and respond to patient deterioration early, thereby reducing complications and improving recovery outcomes.
  Interventions: Behavioral: Risk Early Warning Management
- Routine Perioperative Management: Participants in this arm received standard perioperative care according to hospital guidelines. This included general health education prior to surgery, assistance during the perioperative period, routine postoperative care such as anticoagulation and infection prevention, regular vital signs monitoring, and standard nursing interventions. No specific early warning risk scoring or tiered response strategy was implemented.
  Interventions: Behavioral: Standard Perioperative Care

INTERVENTIONS:
Behavioral: Risk Early Warning Management — This intervention involves a perioperative risk early warning management strategy for hip fracture patients. A dedicated team of nurses is responsible for monitoring vital signs (heart rate, blood pressure, respiratory rate, temperature, and consciousness level) to identify and respond to early signs of clinical deterioration.
  The intervention follows a structured scoring system that classifies patients into different risk levels based on their vital signs:
  Risk Score 0-4: Standard perioperative care and monitoring
  Risk Score 5-7 (or single-item score ≥3): Intensive monitoring with vital sign checks every 4 hours and immediate physician notification if condition changes
  Risk Score ≥7: Continuous monitoring, with immediate physician availability and ready access to emergency equipment The intervention aims to improve patient outcomes by ensuring early identification of deterioration and more rapid response to clinical changes. A red warning sign will also be placed at the patient's b
  Groups: Risk Early Warning Perioperative Management
Behavioral: Standard Perioperative Care — This is the standard care protocol for patients undergoing hip fracture surgery at the study hospital. It includes health education before surgery, regular vital sign monitoring, routine anticoagulation, and infection control management.
  Patients will receive standard perioperative management, including preoperative counseling, assistance with rehabilitation exercises, and monitoring of clinical symptoms and vital signs throughout the surgical and recovery process.
  There is no specific risk early warning scoring system in this group, and intervention is based on routine clinical monitoring.
  Groups: Routine Perioperative Management

SUMMARY:
This clinical study aims to evaluate the effectiveness of a perioperative risk early warning management strategy in patients undergoing surgical treatment for hip fractures. Hip fractures are common in elderly individuals and are associated with a high risk of postoperative complications. Traditional perioperative care may not sufficiently identify and respond to early signs of clinical deterioration.

In this study, patients with hip fractures admitted to the orthopedic department of a single hospital from January 2023 to December 2023 were divided into two groups based on their admission time. Patients admitted between June and December 2023 received the early warning risk management intervention (experimental group), while those admitted between January and May 2023 received routine perioperative care (control group). The early warning management system involved a scoring-based approach using vital signs such as heart rate, respiratory rate, blood pressure, body temperature, and consciousness level to classify patients' risk levels. Nursing staff responded with graded interventions, including enhanced monitoring and rapid physician notification for higher-risk patients.

The study retrospectively enrolled 284 patients in total, with 142 in each group. The primary outcomes include changes in coagulation function, self-care ability (measured by the Exercise of Self-care Agency Scale, ESCA), and hip joint functional recovery (measured by the Hospital for Special Surgery, HSS, score). Secondary outcomes include patient satisfaction and incidence of postoperative complications.

The central hypothesis is that perioperative risk early warning management will improve patient safety, enhance self-care capacity, reduce complications, and promote better recovery outcomes compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unilateral intertrochanteric fracture of the femur confirmed by imaging.
* Age 18 years or older.
* Met the indications for surgical treatment and underwent fracture surgery in the study hospital.
* Stable vital signs and clear consciousness postoperatively.

Exclusion Criteria:

* Presence of hematologic diseases such as coagulation dysfunction.
* Existing lower limb disability, invasive trauma, or other comorbid lesions.
* History of mental disorders, cognitive impairment, or poor compliance with treatment protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study includes adult patients (aged ≥18 years) undergoing PFN fixation for hip fractures at Shiyan People's Hospital (January 2023-December 2023).
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Prothrombin Time (PT) | Preoperative baseline and Postoperative 3 days
  Prothrombin Time (PT) will be measured in seconds using a standardized coagulation analyzer to evaluate the extrinsic coagulation pathway. Preoperative and postoperative PT values will be compared between the intervention and control groups.
Change in Activated Partial Thromboplastin Time (APTT) | Preoperative baseline and Postoperative 3 days
  Activated Partial Thromboplastin Time (APTT) will be measured in seconds to assess the intrinsic coagulation pathway. Preoperative and postoperative APTT values will be compared between groups.
Change in Fibrinogen (FBG) Levels | Preoperative baseline and Postoperative 3 days
  Fibrinogen levels (g/L) will be quantified to reflect clotting factor concentration. Preoperative and postoperative FBG values will be compared between groups.
Change in D-Dimer (D-D) Levels | Preoperative baseline and Postoperative 3 days
  D-dimer levels (mg/L) will be measured to evaluate fibrinolysis activity. Preoperative and postoperative D-D values will be compared between groups.

SECONDARY OUTCOMES:
Change in Exercise of Self-Care Agency Scale (ESCA) Score | Baseline (pre-intervention) and immediately after the intervention
  The ESCA scale evaluates patients' self-care ability across four domains: self-concept, self-responsibility, self-care skills, and health knowledge. Scores range from low to high, with higher scores indicating better self-care agency. Scores will be compared before and after the intervention in each group.
Incidence of Postoperative Complications | Perioperative period to 30 days after Endpoint (day of discharge)
  Complications such as infection, thrombosis, delayed wound healing, and bleeding events will be monitored and recorded. The incidence rate will be compared between the intervention and control groups.
Patient Satisfaction Rate | Immediately after the intervention
  A satisfaction questionnaire will be administered to patients upon discharge. Responses will be categorized as satisfied, neutral, or dissatisfied. The satisfaction rate is calculated as: (satisfied cases / total cases) × 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Shiyan People's Hospital (People's Hospital Affiliated to Hubei Medical College), Shiyan, China

IPD SHARING:
Plan to Share IPD: No